CLINICAL TRIAL: NCT01433198
Title: Aquatic Training in Patients With Severe Scarring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: finances and feasibility
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. Eric Van den Kerckhove, PhD - PT, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML7560
Record Dates: First submitted 2011-09-01; First posted 2011-09-13 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2020-11

CONDITIONS: Burns; Scar
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic exercise group (Active Comparator)
  Interventions: Other: Aquatic training
- Control group (No Intervention)

INTERVENTIONS:
Other: Aquatic training — Aquatic training during a 6 weeks program (15 to 18 sessions of 1 hour)
  Arms: Aquatic exercise group

SUMMARY:
Aim:

- to investigate the effects of an aquatic exercise program in patients with severe scars

Patient population:

* 10 patients of at least 18 years old
* patients with scars after burns or other severe skin injuries
* stratification into two groups: an intervention group and a control group

Method:

* 8 patients will participate in the aquatic exercise group and 2 patients in the control group
* assessment of physical fitness parameters, scar tissue and psychosocial impact

Hypothesis:

- patients of the aquatic exercise group will recover sooner and better (physically and psychologically) than patients of the control group

DETAILED DESCRIPTION:
Intervention:

- during 6 weeks patients will performed an aquatic exercise program (2 to 3 sessions a week)

Assessment:

* T0: post-hospitalisation status: body mass index, physical fitness, strength and respiratory function
* T1: at baseline: body mass index, physical fitness, strength, respiratory function, exercise capacity, mobility, scar parameters and some questionnaires
* T2: after 6 weeks training: same measurements as T1
* T3: 3 months after end of aquatic training: idem T1
* T4: 6 months after end of aquatic training: questionnaires
* T5: 1 year after end of aquatic training: questionnaires

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* hospitalisation at the burn unit of at least 14 days
* patients with severe skin damage (like burns, deglovements, necrotic fasciitis, ...)

Exclusion Criteria:

* younger than 18 years
* psychiatric history (recommandation of psychiatrist not to participate in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity using Dynaport activity monitor | Post-hospitalisation status, baseline, after 6 weeks, after 3 months
  Post-hospitalisation status = participants will be followed during the last three consecutive days of their hospital stay.
  The minimum period of hospital stay is 14 days (inclusion criteria), the maximum period of hospital stay is not determined. The expected average can not be given.

SECONDARY OUTCOMES:
Strength (Jamar, MicroFET, MIP) | Post-hospitalisation status, basline, after 6 weeks, after 3 months
  Strength (Jamar, MicroFET, MIP)
Quality of life (using 5 questionnaires like SF-36) | Basline, after 6 weeks, after 3 months
  Quality of life (using 5 questionnaires like SF-36)
Exercise capacity (6-minutes walking test and 4-minutes swimming test) | Baseline, after 6 weeks and after 3 months
  Exercise capacity (6-minutes walking test and 4-minutes swimming test)
BMI | Post-hospitalisation status, baseline, after 6 weeks and after 3 months
  BMI
Joint mobility | Baseline, after 6 weeks, after 3 months
  Joint mobility
Pulmonary function (FEV1 and FVC) | Post-hospitalisation status, baseline, after 6 weeks, after 3 months
  Pulmonary function (FEV1 and FVC)
Scar assessment | Baseline, after 6 weeks, after 3 months
  Scar assessment
Physical fitness using Squash questionnaire | Baseline, after 6 weeks, after 3 months, after 6 months, after 1 year
  Physical fitness using Squash questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van den Kerckhove, Principal Investigator — KU Leuven